CLINICAL TRIAL: NCT00879892
Title: Phase 2 Study of Effect of Xenon, in Combination With Therapeutic Hypothermia, on the Brain and on Neurological Outcome Following Brain Ischemia in Cardiac Arrest Patients
Brief Title: Effect of Xenon and Therapeutic Hypothermia, on the Brain and on Neurological Outcome Following Brain Ischemia in Cardiac Arrest Patients
Acronym: Xe-hypotheca
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Academy of Finland (Other); University of Turku (Other)
Responsible Party: Principal Investigator, Timo Laitio, Principal investigator, study group leader, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eudra CT2009-009505-25
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Ischemic Brain Injury
Keywords: xenon; hypothermia; out-of-hospital cardiac arrest
MeSH Terms: conditions — Hypothermia; Out-of-Hospital Cardiac Arrest | interventions — Xenon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypothermia and xenon (Active Comparator)
  Interventions: Drug: xenon; Other: Hypothermia
- Hypothermia (Active Comparator)
  Interventions: Other: Hypothermia

INTERVENTIONS:
Drug: xenon — Gas, 24 hour inhalation, en tidal target concentration 40%
  Arms: Hypothermia and xenon
Other: Hypothermia — 24 hour, target core temperature 33

SUMMARY:
The main purpose of this study is to explore whether xenon is neuroprotective in humans. In addition, the purpose is to explore the underlying mechanisms for the possible synergistic neuroprotective interaction of xenon and hypothermia in patients suffering cerebral ischemia post cardiac arrest, by undertaking brain imaging to evaluate their effects on cerebral hypoxia, neuronal loss and mitochondrial dysfunction. In addition, the investigators aim to correlate these findings with neurological outcome to determine surrogate markers of favourable clinical outcome at six months.

DETAILED DESCRIPTION:
If cardiac resuscitation is successful, the state-of-the-art management is to actively cool these patients into a state of moderate hypothermia (32-34º C) for 24 hours in an intensive care unit. Guidelines regarding the use of hypothermia following witnessed cardiac arrest have been formally adopted by the European Resuscitation Council as well as the American Heart Association. Therapeutic hypothermia provides a significant but moderate improvement in these patients. Thus, strategies designed to increase the efficacy of therapeutic hypothermia are needed.

Preclinical animal studies have now demonstrated a remarkable neuroprotective interaction with hypothermia in a synergistic manner. The data suggest that xenon's neuroprotective effect can be triggered with subanesthetic concentrations in humans when combined with modest hypothermia.

The aim of this study is to explore whether xenon is neuroprotective in humans. We also explore whether xenon in combination with standard hypothermia treatment has better neuroprotective effect than can be achieved with the hypothermia treatment alone in the patients who have experienced global ischemic brain injury after out-of-hospital cardiac arrest (OHCA).

Hundred-and- ten patients who have experienced ventricular fibrillation or non-perfusive ventricular tachycardia as initial cardiac rhythm will be enrolled and they will be randomized into two treatment groups: 1) standard hypothermia treatment for 24 hours, 2) xenon inhalation combined with standard hypothermia treatment for 24 hours.

Sophisticated brain imaging techniques will be performed before intervention (i.e. standard CT scan), within 24 hours after intervention (i.e. positron emission tomography), and on day 3 and on day 10 after cardiac arrest (i.e. various proton magnetic resonance imaging techniques) to identify ischemic burden, injured tissue and deranged energy metabolism in the brain.

Our objective is to show a significant reduction in the degree of severity of the ischemic brain injury in the hypothermia+Xenon group as compared with the hypothermia group.

ELIGIBILITY:
Inclusion Criteria:

1. Ventricular fibrillation or non-perfusive ventricular tachycardia as initial cardiac rhythm
2. The 1st attempt at resuscitation by emergency medical personnel must appear within 15 minutes after the collapse
3. The cause for collapse should be considered primary as cardiogenic and the return of spontaneous circulation (ROSC) should have been gained in 45 minutes after the collapse
4. Patient should be still unconscious in the emergency room
5. Age: 18 - 80 years
6. Obtained consent within 4 hours after arrival to the hospital

Exclusion criteria

1. Hypothermia (< 30°C core temperature)
2. Unconsciousness before cardiac arrest (cerebral trauma, spontaneous cerebral hemorrhages, intoxications etc.)
3. Response to verbal commands after the return of spontaneous circulation and before randomization
4. Pregnancy
5. Coagulopathy
6. Terminal phase of a chronic disease
7. Systolic arterial pressure < 80 mmHg or mean arterial pressure < 60 mmHg for over 30 min period after ROSC
8. Evidence of hypoxemia (arterial oxygen saturation < 85%) for > 15 minutes after ROSC and before randomization.
9. Factors making participation in follow-up unlikely
10. Enrolment in another study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2009-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome is to show a significant reduction in the degree of severity of the ischemic brain injury in the hypothermia+Xenon group as compared with the hypothermia group, reflected by various MRI techniques | within 24 hours after treatment and 10 +/-2 days after cardiac arrest
  Power analysis was done with fractional anisotropy of diffusion tensor MRI

SECONDARY OUTCOMES:
Neurological outcome | 6 months after cardiac arrest
A transthoracic echocardiography will be performed for all feasible patients to investigate cardiac safety of the treatments | Before, during and after treatments
Mortality | 6 months
Complication rate | 7 days
  epileptic status, severe bleeding, pneumonia, sepsis, pancreatitis, acute kidney injury according to RIFLE, pulmonary oedema, arrhythmias
Morbidity | 6 months
  cardiac and cerebral morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Timo T Laitio, MD, PhD, Principal Investigator — Department of Anaesthesiology, Intensive Care, Emergency Care and Pain Medicine
Locations (10):
- Department of Anesthesia and Perioperative Care, San Francisco, California, United States
- Finland (9):
  - Department of Neurology, Meilahti, Helsinki University Hospital, Helsinki
  - Department of Radiology, HUSRontgen, Meilahti, Helsinki University Hospital, Helsinki
  - Intensive Care Unit, Meilahti, Helsinki University Hospital, Helsinki
  - Department of Cardiology, Meilahti, Helsinki University Hospital, Helsinki
  - Adult Intensive Care Unit, Turku University Hospital, Turku
  - Department of Internal Medicine, Division of Cardiology, Turku University Hospital, Turku
  - Department of Neurology; Turku University Hospital, Turku
  - Department of Radiology, Turku University Hospital, Turku
  - PET Centre, Turku

REFERENCES:
- [Background] Hypothermia after Cardiac Arrest Study Group. Mild therapeutic hypothermia to improve the neurologic outcome after cardiac arrest. N Engl J Med. 2002 Feb 21;346(8):549-56. doi: 10.1056/NEJMoa012689. PMID 11856793
- [Derived] Hollmen CC, Vorobyev V, Parkkola R, Posti JP, Saunavaara J, Laitio R, Arola O, Hynninen M, Backlund M, Blennow K, Zetterberg H, Martola J, Ylikoski E, Roine RO, Tiainen M, Scheinin H, Maze M, Vahlberg T, Laitio TT; Xe-HYPOTHECA Consortium. Grey matter volume reduction and its association with brain-enriched blood biomarkers in out-of-hospital cardiac arrest survivors. Sci Rep. 2025 Nov 26;15(1):42219. doi: 10.1038/s41598-025-26322-4. PMID 41298726
- [Derived] Hollmen C, Parkkola R, Vorobyev V, Saunavaara J, Laitio R, Arola O, Hynninen M, Backlund M, Martola J, Ylikoski E, Roine RO, Tiainen M, Scheinin H, Maze M, Vahlberg T, Laitio TT. Neuroprotective Effects of Inhaled Xenon Gas on Brain Structural Gray Matter Changes After Out-of-Hospital Cardiac Arrest Evaluated by Morphometric Analysis: A Substudy of the Randomized Xe-Hypotheca Trial. Neurocrit Care. 2025 Feb;42(1):131-141. doi: 10.1007/s12028-024-02053-8. Epub 2024 Jul 9. PMID 38982000
- [Derived] Nummela AJ, Scheinin H, Perola M, Joensuu A, Laitio R, Arola O, Gronlund J, Roine RO, Backlund M, Vahlberg TJ, Laitio T; Xe-Hypotheca Collaboration Group. A metabolic profile of xenon and metabolite associations with 6-month mortality after out-of-hospital cardiac arrest: A post-hoc study of the randomised Xe-Hypotheca trial. PLoS One. 2024 Jun 4;19(6):e0304966. doi: 10.1371/journal.pone.0304966. eCollection 2024. PMID 38833442
- [Derived] Koskensalo K, Virtanen S, Saunavaara J, Parkkola R, Laitio R, Arola O, Hynninen M, Silvasti P, Nukarinen E, Martola J, Silvennoinen HM, Tiainen M, Roine RO, Scheinin H, Saraste A, Maze M, Vahlberg T, Laitio TT; XeHYPOTHECA Research Group. Comparison of the prognostic value of early-phase proton magnetic resonance spectroscopy and diffusion tensor imaging with serum neuron-specific enolase at 72 h in comatose survivors of out-of-hospital cardiac arrest-a substudy of the XeHypotheca trial. Neuroradiology. 2023 Feb;65(2):349-360. doi: 10.1007/s00234-022-03063-z. Epub 2022 Oct 17. PMID 36251060
- [Derived] Laitio R, Hynninen M, Arola O, Virtanen S, Parkkola R, Saunavaara J, Roine RO, Gronlund J, Ylikoski E, Wennervirta J, Backlund M, Silvasti P, Nukarinen E, Tiainen M, Saraste A, Pietila M, Airaksinen J, Valanne L, Martola J, Silvennoinen H, Scheinin H, Harjola VP, Niiranen J, Korpi K, Varpula M, Inkinen O, Olkkola KT, Maze M, Vahlberg T, Laitio T. Effect of Inhaled Xenon on Cerebral White Matter Damage in Comatose Survivors of Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2016 Mar 15;315(11):1120-8. doi: 10.1001/jama.2016.1933. PMID 26978207
- [Derived] Arola OJ, Laitio RM, Roine RO, Gronlund J, Saraste A, Pietila M, Airaksinen J, Perttila J, Scheinin H, Olkkola KT, Maze M, Laitio TT. Feasibility and cardiac safety of inhaled xenon in combination with therapeutic hypothermia following out-of-hospital cardiac arrest. Crit Care Med. 2013 Sep;41(9):2116-24. doi: 10.1097/CCM.0b013e31828a4337. PMID 23896830